CLINICAL TRIAL: NCT01046058
Title: A Phase I, Open-label, Sequential Trial to Investigate the Pharmacokinetics, Safety, and Tolerability of TMC435 in Subjects With Moderately or Severely Impaired Hepatic Function
Brief Title: TMC435-TiDP16-C113: A Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics of TMC435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016783; TMC435-TiDP16-C113 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hepatitis C Virus
Keywords: TMC435-TiDP16-C113; TMC435-C113; TMC435; HCV; Protease Inhibitor; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panel A: TMC435 150 mg (Experimental): Participants enrolled in Panel A had moderate hepatic failure and received TMC435 150 mg once daily for 7 days.
  Interventions: Drug: TMC435
- Panel B: TMC435 150 mg (Experimental): Participants enrolled in Panel B had severe hepatic impairment and received TMC435 150 mg once daily for 7 days after the safety of TMC435 150 mg once daily for 7 days was evaluated in participants enrolled in Panel A.
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — 150 mg (two 75-mg capsules) orally (by mouth) once daily for 7 days

SUMMARY:
The purpose of the study is to investigate the effect of moderate and severe hepatic impairment on the pharmacokinetics of TMC435. Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. In addition, the short-term safety and tolerability of TMC435 in participants with hepatic impairment will be determined. The results of this study will guide dose recommendations for TMC435 in patients with impaired liver function.

DETAILED DESCRIPTION:
This is a Phase I, open-label trial to investigate the pharmacokinetics (how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body) of TMC435 in 8 participants with moderate hepatic impairment and 8 participants with severe hepatic impairment as compared to 8 participants with normal hepatic function, matched for age, gender, race, BMI (body mass index = weight in kilogram divided by square of height in meters) and smoking status. Open-label means that the study doctor and the participants know what treatment will be assigned to them. All participants will receive 150 mg of TMC435 by mouth for 7 days. Participants with severe hepatic impairment will be treated when the pharmacokinetic profiles of TMC435 in participants with moderate hepatic impairment have been evaluated. The dose of TMC435 may be changed for participants with severe hepatic impairment after evaluation of the blood levels TMC435 in participants with moderately impaired hepatic function. Tolerability and safety of TMC435 will be assessed throughout the trial period. Illnesses and side effects will be checked at every visit. Blood samples will be taken at screening, on the day before TMC435 intake, on days 2, 3, 5, 6, 7 (11 times), 8 and 9 and at 2 follow-up visits. Blood levels of TMC435 will be determined on days 2, 5, 6, 7, 8 and 9. Urine samples, ECG and vital signs will be taken at screening, twice on day 7 and at 2 follow-up visits. A physical examination will be done at screening, on the day before TMC435 intake, on day 9 and at both follow-up visits. All participants will receive a 150 mg dose of TMC435 for 7 days, given by mouth as 2 capsules of 75 mg. After evaluation of the pharmacokinetic profiles of TMC435 in participants with moderate hepatic impairment, the dose may be changed for participants with severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hepatic impairment: Moderate or severe hepatic impairment, clinically diagnosed as Child Pugh B or C
* Stable liver cirrhosis and hepatic impairment for at least 3 months prior to the start of the study. Participants with normal hepatic function: Healthy based on a medical evaluation including medical history, physical examination, blood tests and electrocardiogram

Exclusion Criteria:

* Participants with hepatic impairment: Fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment within 3 months prior or within the screening period
* Cirrhosis due to chronic hepatitis B or C infection. Participants with normal hepatic function: History or presence of hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of TMC435 in patients with moderate and severe hepatic impairment | Measured at 16 predefined time points over a period of 9 days. Extensive analysis is planned on Day7 (after last intake of TMC435), with 12 PK sampling moments over 48 hours.

SECONDARY OUTCOMES:
Short-term safety and tolerability of TMC435 in volunteers with moderate or severe hepatic impairment | AEs monitored each visit; vital signs, urinalysis and ECG parameters on Day 7 and on both follow-up visits; Safety blood sample at 6 predefined timepoints (over 5 days) and on both follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (3):
- United States (3):
  - Anaheim, California
  - Orlando, Florida
  - San Antonio, Texas

REFERENCES:
- See also: A Phase I, open-label, sequential trial to investigate the pharmacokinetics, safety, and tolerability of TMC435 in subjects with moderately or severely impaired hepatic function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1034&filename=CR016783_CSR.pdf